CLINICAL TRIAL: NCT02699047
Title: Gastrointestinal Cancer: Effects of the Fish Oil Intake on Nutritional Status, Quality of Life and Immune and Metabolic Outcomes
Brief Title: Fish Oil Supplementation in Gastrointestinal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal de Santa Catarina (Other)
Collaborators: Centro de Pesquisas Oncológicas (Other)
Responsible Party: Principal Investigator, Erasmo Benicio Santos de Moraes Trindade, Ph.D. Professor, Universidade Federal de Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UFSC/04
Record Dates: First submitted 2016-02-12; First posted 2016-03-04 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Gastrointestinal Cancer; Colorectal Cancer; Stomach Cancer
Keywords: Gastrointestinal cancer; Fish oil; Oxidative stress; Inflammation; Quality of life; Nutritional status; Colorectal cancer; Stomach cancer; Chemotherapy; polyunsaturated fatty acids n-3
MeSH Terms: conditions — Gastrointestinal Neoplasms; Colorectal Neoplasms; Stomach Neoplasms; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fish oil (Experimental): 3.6 g/day of the encapsulated fish oil (2 capsules/day) providing 1.55 g/d of the n-3 polyunsaturated fatty acids (EPA and DHA) during 9 weeks
  Interventions: Dietary Supplement: Encapsuled fish oil
- Control group (Placebo Comparator): 3.2 g/day of the olive oil (2 capsules/day) without n-3 polyunsaturated fatty acids
  Interventions: Dietary Supplement: Encapsulated Olive oil

INTERVENTIONS:
Dietary Supplement: Encapsuled fish oil — Fish oil extracted from sardine, mackerel and anchovy. Nutritional information per capsule: Kcal: 13; protein: 0.35g; Total Fats: 1.25g; Saturated fat: 0g; polyunsaturated fat: 0.75g; EPA: 0.5g; DHA: 0.25g; Cholesterol: 0g. The supplement was provided in gelatinous capsule with antioxidant (tocopherols).
  Arms: Fish oil
Dietary Supplement: Encapsulated Olive oil — Extra virgin olive oil. Nutritional information per capsule: Kcal: 10; protein: 0.35g; Total Fats: 1g; Saturated fat: 0.1 g; monounsaturated fat: 0.75g; polyunsaturated fat: 0.1g; EPA: 0g; DHA: 0g; oleic acid: 0.65g; Cholesterol: 0g. The supplement was provided in gelatinous capsule without antioxidants.
  Arms: Control group

SUMMARY:
Double-blind, randomized clinical trial to assess the effects of 1,55 g/day of n-3 fatty acids from fish oil concomitant chemotherapy in gastrointestinal cancer.

DETAILED DESCRIPTION:
This study will be divided into three stages defined as: baseline (T0), middle moment (T1) and final moment (T2). At baseline, will be performer the patients identification, clinical data collection, assessment of anthropometric data and body composition, blood sample collection and questionnaires application for individuals allocated into two groups (Fish Oil Group and Placebo Group). The Fish Oil Group (GOP) will receive fish oil capsules and the placebo group (GP) will receive capsules containing olive oil, both also will receive consumption guidelines.

The list of randomization was generated by a computer program and was divided by cancer localization and gender. The researchers involved with the recruitment had access only to randomization list containing codes. The codes were distributed sequentially.

The baseline is the day of first chemotherapy. In the middle moment, five weeks after the start of study, new blood collection, questionnaires and measurement of anthropometric data will be performed. At the final moment, nine weeks after baseline, last blood collection, questionnaires and measurement of anthropometric data and body composition of fish oil and placebo groups will be performed, and will feature the end of the capsules consumption.

After 6 months and 1 year after the initiation of chemotherapy and supplementation with fish oil or placebo, survival data will be collected.

Throughout the monitoring period, the researcher and collaborators will maintain contact with the individuals included. The contact will be made in CEPON, where they receive chemotherapy, and by telephone.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with age between 18 to 70 y.
* Histopathological diagnosis of gastric cancer, or colorectal or anal canal or intestinal cancer
* Ability to start chemotherapy in institution (CEPON)
* Performance status <= 2

Exclusion Criteria:

* Prior chemotherapy
* Inability to oral intake
* diagnosis of infectious or inflammatory disease or diabetes
* Allergy to fish and / or derivatives,
* Pregnant,
* Treatment with statins or anti-inflammatories drugs
* Intake of fish oil and/or another supplement containing omega-3 or other polyunsaturated fatty acid in the six months prior their inclusion in the study
* Continued use of supplements containing antioxidants
* Patients in palliative care
* without cognitive ability to perform the study protocol
* Enrolled in studies with new drugs
* Hospitalized patients at recruitment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-03; Primary Completion 2016-04 (Actual); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of life | baseline and 9 weeks (final moment)
  Application by interview of the EORTC QOL questionnaires: QLQ-C30 v. 3.0; CRC-29 and STO22. The change was observed by increase ou decrease in overall score of the scales.
Cytokines of inflammatory response | Baseline, 5 and 9 weeks
  Quantification of plasmatic concentration of cytokines (TNF, IL-17A, IL-10)
Body weight | 5 and 9 weeks
  Assessment of weight (kg)
Body Mass Index (BMI) | baseline, 5 and 9 weeks
  Assessment of BMI (Kg/m²)
Weight Change | baseline, 5 and 9 weeks
  Weight change in comparison with the weight at baseline (Kg)
Fat mass | baseline and 9 weeks
  Fat mass assessment by electric bioimpedance (kg and %)
Lean body mass | baseline and 9 weeks
  Lean body mass assessment by electric bioimpedance (kg and %)
arm circumference | baseline, 5 and 9 weeks
  measurement of arm circumference using a inelastic metric tape (cm)
tricipital skinfold | baseline, 5 and 9 weeks
  measurement of triciptal skinfold using a caliper (mm)
Serum C-reactive protein | baseline, 5 and 9 weeks
  Serum quantification of C-reactive protein (mg/dL)
Activity of Catalase | Baseline and 9 weeks
  Quantification of erythrocyte catalase activity
Activity of Glutathione Peroxidase | Baseline and 9 weeks
  Quantification of erythrocyte glutathione peroxidase activity
Activity of Superoxide Dismutase | Baseline and 9 weeks
  Quantification of erythrocyte superoxide dismutase activity
Lipid Peroxidation | Baseline and 9 weeks
  Evaluation of lipid hydroperoxides in plasma and leukocytes
Evaluation of adverse events consequences | Baseline and 9 weeks
  Evaluation of changes in treatment protocol due to adverse events (hospitalizations, treatment interruption, delay of treatment administration, dose reductions)
Graduation of adverse events | Baseline, 5 weeks and 9 weeks
  Graduation of hematological and gastrointestinal adverse events related to chemotherapy treatment
Tumor Markers | Baseline and 9 weeks
  Quantification of serum tumor marker CEA and CA19
Survival | Baseline, 6 months and one year
  Evaluation of survival after 6 months and after one year of recruitment
Serum albumin | baseline, 5 weeks and 9 weeks
  Serum quantification of albumin (g/dL)

CONTACTS AND LOCATIONS:
Locations (1):
- Michel Carlos Mocellin, Florianópolis, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Camargo CQ, Mocellin MC, Brunetta HS, Chagas TR, Fabre MES, Trindade EBSM, Silva ELD, Nunes EA. Fish oil decreases the severity of treatment-related adverse events in gastrointestinal cancer patients undergoing chemotherapy: A randomized, placebo-controlled, triple-blind clinical trial. Clin Nutr ESPEN. 2019 Jun;31:61-70. doi: 10.1016/j.clnesp.2019.02.015. Epub 2019 Mar 14. PMID 31060836